CLINICAL TRIAL: NCT04782505
Title: A Open-label, Single-dose, Phase 1 Study to Compare and Evaluate the Safety and Pharmacokinetics According to the Dose of Camostat Mesylate in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Evaluation Study According to the Dose of Camostat Mesylate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1248101
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part1. Parallel, Part2. Crossover
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Part 1) (Experimental): DWJ1248 100mg (100mg 1tab) PO
  Interventions: Drug: DWJ1248
- Cohort 2 (Part 1) (Experimental): DWJ1248 200mg (100mg 2tab) PO
  Interventions: Drug: DWJ1248
- Cohort 3 (Part 1) (Experimental): DWJ1248 300mg (100mg 3tab) PO
  Interventions: Drug: DWJ1248
- Group A (Part 2) (Experimental): DWJ1248 100mg 2tab PO - Wash out - DWJ1248 200mg 1tab PO
  Interventions: Drug: DWJ1248
- Group B (Part 2) (Experimental): DWJ1248 200mg 1tab PO - Wash out - DWJ1248 100mg 2tab PO
  Interventions: Drug: DWJ1248

INTERVENTIONS:
Drug: DWJ1248 — Camostat mesylate Tablet from Daewoong

SUMMARY:
Safety and pharmacokinetics evaluation study according to the dose of camostat mesylate in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 19 and ≤ 55 years at screening
* Subjects with body weight of ≥ 55.0 kg and ≤ 90.0 kg, and a body mass index (BMI) of ≥ 18.0 and ≤ 29.9
* Subjects who have no congenital or chronic disease and have no pathological symptoms or findings as a result of an internal examination

Exclusion Criteria:

* Subjects with current or prior history of a clinically significant hepatic, renal, nervous, respiratory, gastrointestinal, endocrine, hematologic and oncologic, urogenital, cardiovascular, musculoskeletal or psychiatric disorder
* Subjects with symptoms of acute disease within 28 days prior to the scheduled first administration date of IP
* Subjects with a history of gastrointestinal diseases (e.g., Crohn's disease, ulcers, etc.) or gastrointestinal resection (except simple appendectomy or hernia surgery) that may affect the absorption of drugs.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Cmax of GBPA | 0-6 hr
  Maximum blood concentration of GBPA (GUANIDINO BENZOYLOXY PHENYLACETIC ACID METHANESULFONATE) among observed blood concentrations at time points
  * Immediately before administration of IP
  * After administration
AUClast of GBPA | 0-6 hr
  Area under the blood concentration-time of GBPA (GUANIDINO BENZOYLOXY PHENYLACETIC ACID METHANESULFONATE) among observed blood concentrations at time points
  * Immediately before administration of IP
  * After administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No